CLINICAL TRIAL: NCT06427070
Title: Effectiveness of Two Intracanal Irrigation Solutions Delivered Through Cryotherapy on Post-Endodontic Pain Relieve. A Randomized Clinical Trial
Brief Title: Effectiveness of Two Intracanal Irrigation Solutions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Manal Mohamed, Lecturer at Misr university, Misr University for Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHX 2024
Record Dates: First submitted 2024-05-14; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Irreversible Pulpitis
Keywords: Pulpitis; CHX; Saline
MeSH Terms: conditions — Pulpitis | interventions — dextran - saline drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Irrigating solutions (Experimental): Group 1 sodium hypochlorite Group 2 saline Group 3 chlorohexidine
  Interventions: Other: Irrigating solution

INTERVENTIONS:
Other: Irrigating solution — Saline, sodium hypochlorite, chlorohexidine
  Other Names: Chlorohexidine

SUMMARY:
The aim of the present clinical trial is to investigate and compare the effect of crayotherapy utilizing two intra-canal final irrigating solutions on postoperative pain.

DETAILED DESCRIPTION:
1. st: Comparison of pain reduction algorism after cryotherapy using the two tested irrigating materials
2. nd. Number and frequency of analgesics taken for pain relief during one week postoperative

ELIGIBILITY:
Inclusion Criteria:

* Case diagnosed as having symptomatic irreversible pulpitis with symptomatic apical periodontitis
* Patients requiring emergency RCT
* Pre-operative pain score 7 on Numerical Rating (NRS) scale
* Middle aged males (25-50)
* Medical profile ASA1
* Willing to sign the consent form
* Willing to answer our call for one week period

Exclusion Criteria:

* Females
* Medical conditions above ASA1
* Multi-rooted teeth
* Patients younger or older than (25-50)

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Estimated)
Dates: Start 2024-05-23 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
pain scale | 1 week
  pain scale Comparison of the 2 selected irrigating solutions
Analgesics Frequency | 1 week
  Frequency of analgesics for pain relief